CLINICAL TRIAL: NCT05604430
Title: Pre-hospital Ventilation Clinical Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 76701
Record Dates: First submitted 2022-07-11; First posted 2022-11-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Altered Mental Status; Sepsis; Heart Failure; Hemorrhage; Respiratory Distress Syndrome, Adult; Cardiac Arrest
Keywords: Ventilation; Pre-Hospital
MeSH Terms: conditions — Sepsis; Heart Failure; Hemorrhage; Respiratory Distress Syndrome; Heart Arrest; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Ventilator patients: Patients being ventilated by the ZOLL 731 Series ventilator in accordance with device labeling and Agency protocols in a pre-hospital setting.
  Interventions: Device: 731 Series Ventilator

INTERVENTIONS:
Device: 731 Series Ventilator — FDA cleared ventilator indicated for use in the management of acute or chronic respiratory failure or during resuscitation.

SUMMARY:
This study will collect and characterize ventilator use during patient care with a ZOLL 731 Series ventilator in a pre-hospital setting.

DETAILED DESCRIPTION:
This is a prospective, observational study.

ZOLL will develop a methodology to collect and transfer ventilator data from the device to ZOLL to allow for a characterization of ventilator use in the pre-hospital setting. This knowledge and experience will subsequently be used to inform development of a mechanism to allow for automatic data collection and transmission from ZOLL ventilators to a central data repository. These data will be used to provide feedback, reporting, and benchmarking to individual agencies and departments on their ventilator use as well as aggregate use data from all ventilators to allow for comparisons.

Enrollment in this study is expected to take approximately 24 months. No patient outcome data will be collected.Participants are enrolled once data have been downloaded from the ventilator via RescueNet® VentReview software. Participants will not be followed after the assessment of study objectives.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for this study must meet all of the following Inclusion criteria:

  1. Ventilated using ZOLL 731 Series ventilator with Release 5 (or greater) software
  2. Data recorded in ventilator data file

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cases where participating EMS Agencies use ZOLL 731 Series ventilator in accordance with device labeling and Agency protocols in a pre-hospital setting
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2030-04-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Ventilator modes used | Through study completion, an average 1 hour
  Characterizing how often ventilator modes are used during mechanical ventilation
Ventilator settings used | Through study completion, an average 1 hour
  Characterizing how often ventilator settings are changed during mechanical ventilation
Ventilator Alarm type | Through study completion, an average 1 hour
  Characterize type of alarms triggered during mechanical ventilation
Ventilator Alarm Frequency | Through study completion, an average 1 hour
  Characterize frequency of alarms triggered during mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - East Baton Rouge EMS, Baton Rouge, Louisiana
  - Uxbridge Fire, Uxbridge, Massachusetts
  - MedStar, Fort Worth, Texas
  - Gig Harbor Fire Department, Rosedale, Washington

IPD SHARING:
Plan to Share IPD: No